CLINICAL TRIAL: NCT02074059
Title: A Multicenter, Randomized, Open-Label, Controlled Trial to Assess the Safety and Tolerability of Lucinactant for Inhalation in Preterm Neonates 29 to 34 Weeks PMA: Dose Escalation and Study Extension
Brief Title: Trial to Assess the Safety and Tolerability of Lucinactant for Inhalation in Premature Neonates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 03-CL-1201; 4R44HL107000-02 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — lucinactant; Inhalation; Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Sequential escalating dosing groups, each group contained an active and control arm of equal size.
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Aerosolized lucinactant (25 mg/kg) (Experimental): 25 mg total phospholipids (TPL)/kg: Lucinactant for inhalation with nCPAP
  Interventions: Drug: Lucinactant for Inhalation
- Aerosolized lucinactant (50 mg/kg) (Experimental): 50 mg TPL/kg: Lucinactant for inhalation with nCPAP
  Interventions: Drug: Lucinactant for Inhalation
- Aerosolized lucinactant (75 mg/kg) (Experimental): 75 mg TPL/kg: Lucinactant for inhalation with nCPAP
  Interventions: Drug: Lucinactant for Inhalation
- Aerosolized lucinactant (100 mg/kg) (Experimental): 100 mg TPL/kg: Lucinactant for inhalation with nCPAP; repeat dosing possible if criteria met.
  Interventions: Drug: Lucinactant for Inhalation
- Aerosolized lucinactant (150 mg/kg) (Experimental): 150 mg TPL/kg: Lucinactant for inhalation with nCPAP; repeat dosing possible if criteria met.
  Interventions: Drug: Lucinactant for Inhalation
- nCPAP alone (Active Comparator): nCPAP therapy alone
  Interventions: Device: nCPAP alone

INTERVENTIONS:
Drug: Lucinactant for Inhalation — Lucinactant for Inhalation refers to the active investigational agent, lucinactant, in combination with the investigational delivery device (drug-device combination product)
  Other Names: Aerosurf
  Arms: Aerosolized lucinactant (100 mg/kg); Aerosolized lucinactant (150 mg/kg); Aerosolized lucinactant (25 mg/kg); Aerosolized lucinactant (50 mg/kg); Aerosolized lucinactant (75 mg/kg)
Device: nCPAP alone — nCPAP therapy
  Other Names: nasal continuous positive airway pressure
  Arms: nCPAP alone

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of aerosolized surfactant, specifically lucinactant for inhalation, administered in escalating inhaled doses to preterm neonates 29 to 34 weeks gestational age who are receiving nasal continuous positive airway pressure (nCPAP) for respiratory distress syndrome (RDS), compared to neonates receiving nCPAP alone.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from a legally authorized representative
* Gestational age 29 to 34 completed weeks (34 weeks 6 days) post menstrual age (PMA)
* Successful implementation of controlled nCPAP within 90 minutes after birth
* Spontaneous breathing
* Chest radiograph consistent with RDS
* Need for moderate levels of supplemental oxygen and nCPAP to maintain oxygen saturation of 88% to 95% for at least 30 minutes within the first 21 hours after birth

Exclusion Criteria:

* Heart rate that cannot be stabilized above 100 beats/minute within 5 minutes of birth
* Recurrent episodes of apnea occurring after the initial newborn resuscitation period (ie, 10 minutes after birth) requiring intermittent positive pressure breaths using inflating pressures above the set CPAP pressure administered manually or mechanically through any patient interface
* A 5 minute Apgar score < 5
* Major congenital malformation(s) and cranial/facial abnormalities that preclude nCPAP, diagnosed antenatally or immediately after birth
* Other diseases or conditions potentially interfering with cardiopulmonary function (eg, hydrops fetalis or congenital infection such as TORCH)
* Known or suspected chromosomal abnormality or syndrome
* Prolong rupture of membranes (PROM) > 2 weeks
* Evidence of hemodynamic instability requiring vasopressors or steroids for hemodynamic support and/or presumed clinical sepsis
* Need for endotracheal intubation and mechanical ventilation
* Has been administered: another investigational agent or exposure to an investigational medical device, any other surfactant agent, steroid treatment after birth

Ages: 29 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Segal, MD, FACP, Principal Investigator — Windtree Therapeutics, Inc.
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Christiana Care Health System, Newark, Delaware
  - University of Miami, Miami, Florida
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Mid Atlantic Neonatology Associates, Morristown, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Providence St. Vincent Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerolized Lucinactant (25 mg/kg): 25 mg TPL/kg of Lucinactant for inhalation with nCPAP
- Aerosolized Lucinactant (50 mg/kg): 50 mg TPL/kg of Lucinactant for inhalation with nCPAP
- Aerosolized Lucinactant (75 mg/kg): 75 mg TPL/kg of Lucinactant for inhalation with nCPAP
- Aerosolized Lucinactant (100 mg/kg): 100 mg TPL/kg of Lucinactant for inhalation with nCPAP; 1 repeat dose allowed if repeat dosing criteria were met
- Aerosolized Lucinactant (150 mg/kg): 150 mg TPL/kg of Lucinactant for inhalation with nCPAP; 1 repeat dose allowed if repeat dosing criteria were met
Period: Overall Study
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (75 mg/kg) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone
Started | 8 | 8 | 8 | 8 | 8 | 40
Completed | 8 | 8 | 8 | 8 | 7 | 39
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (75 mg/kg) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 8 | 8 | 8 | 40 | 80
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 3 | 6 | 21 | 42
  Male | 5 | 3 | 4 | 5 | 2 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 2 | 2 | 2 | 11 | 22
  Not Hispanic or Latino | 7 | 4 | 6 | 6 | 6 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 0 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 0 | 4 | 7
  White | 4 | 5 | 4 | 5 | 6 | 30 | 54
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 1 | 2 | 2 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 40 | 80
Gestational Age [Mean (Standard Deviation); unit: weeks] | 30.5 (0.81) | 31.8 (1.50) | 33.3 (2.11) | 31.7 (2.10) | 32.3 (1.95) | 31.5 (1.56) | 31.7 (1.74)

OUTCOME MEASURES:

1. Primary Outcome: Peri-Dosing Events
Description: Pre-specified adverse events that occured during treatment administration; does not include nCPAP alone
Time Frame: Within 48 Hours after Initiation of Study Treatment
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (75 mg/kg) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 0
participants
  Bradycardia | 0 | 0 | 0 | 1 | 0 |
  Desaturation | 2 | 0 | 1 | 2 | 0 |
  Vomiting | 0 | 0 | 1 | 1 | 0 |

2. Primary Outcome: All Cause Mortality
Time Frame: Within 36 Weeks PMA
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (75 mg/kg) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
participants | 0 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Oxygen Saturation Levels
Description: Oxygen saturation as determined by pulse oximetry
Time Frame: Within 3 Hours of Randomization
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (75 mg/kg) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
percentage of oxygen saturation
  At Randomization: number analyzed (Participants) | 1 | 6 | 8 | 8 | 8 | 30
  At Randomization | 94.0 (0) | 91.3 (2.73) | 96.4 (2.20) | 93.9 (3.87) | 92.5 (3.85) | 93.3 (2.66)
  At Initiation of Treatment: number analyzed (Participants) | 4 | 6 | 7 | 8 | 8 | 0
  At Initiation of Treatment | 93.0 (4.00) | 93.3 (1.37) | 93.4 (4.24) | 94.0 (3.82) | 93.1 (1.25) |
  15 Minutes Post Radomization/Treatment: number analyzed (Participants) | 1 | 6 | 8 | 8 | 8 | 36
  15 Minutes Post Radomization/Treatment | 94.0 (0) | 92.7 (4.68) | 94.8 (5.15) | 94.8 (3.62) | 92.0 (4.66) | 93.3 (3.39)
  30 Minutes Post Randomization/Treatment: number analyzed (Participants) | 2 | 6 | 8 | 8 | 8 | 32
  30 Minutes Post Randomization/Treatment | 93.5 (2.12) | 92.3 (2.25) | 92.5 (5.95) | 93.3 (4.83) | 91.4 (3.89) | 93.6 (3.33)
  45 Minutes Post Randomization/Treatment: number analyzed (Participants) | 2 | 6 | 8 | 8 | 8 | 31
  45 Minutes Post Randomization/Treatment | 94.5 (0.71) | 91.3 (3.88) | 94.0 (4.72) | 93.8 (3.11) | 93.0 (2.27) | 93.7 (3.04)
  60 Minutes Post Randomization/Treatment: number analyzed (Participants) | 1 | 6 | 8 | 8 | 8 | 33
  60 Minutes Post Randomization/Treatment | 92.0 (0) | 93.7 (2.07) | 96.1 (2.47) | 93.9 (3.72) | 91.9 (3.00) | 93.5 (3.68)
  1.25 Hours Post Randomization/Treatment: number analyzed (Participants) | 1 | 6 | 8 | 7 | 8 | 31
  1.25 Hours Post Randomization/Treatment | 94.0 (0) | 93.2 (4.71) | 95.6 (2.33) | 94.0 (3.32) | 92.0 (5.26) | 93.9 (3.05)
  1.5 Hours Post Randomization/Treatment: number analyzed (Participants) | 2 | 6 | 8 | 7 | 8 | 32
  1.5 Hours Post Randomization/Treatment | 95.0 (4.24) | 93.7 (3.27) | 94.9 (3.52) | 93.1 (6.34) | 88.1 (16.98) | 93.4 (2.83)
  1.75 Hours Post Randomization/Treatment: number analyzed (Participants) | 3 | 6 | 8 | 7 | 8 | 30
  1.75 Hours Post Randomization/Treatment | 92.3 (8.33) | 93.3 (4.13) | 95.4 (2.45) | 94.6 (4.72) | 93.4 (5.42) | 93.9 (2.61)
  2.00 Hours Post Radomization/Treatment: number analyzed (Participants) | 1 | 6 | 8 | 8 | 8 | 30
  2.00 Hours Post Radomization/Treatment | 97.0 (0) | 90.2 (6.24) | 95.0 (2.78) | 93.9 (3.87) | 93.4 (3.58) | 93.5 (2.33)
  2.25 Hours Post Randomization/Treatment: number analyzed (Participants) | 2 | 6 | 8 | 7 | 8 | 30
  2.25 Hours Post Randomization/Treatment | 90.5 (2.12) | 92.3 (2.42) | 94.5 (3.38) | 94.9 (3.18) | 92.8 (4.46) | 93.4 (2.63)
  2.50 Hours Post Randomization: number analyzed (Participants) | 1 | 6 | 8 | 7 | 8 | 31
  2.50 Hours Post Randomization | 91.0 (0) | 93.3 (1.37) | 95.0 (2.62) | 94.0 (3.61) | 93.6 (4.31) | 93.4 (3.19)
  2.75 Hours Post Randomization/Treatment: number analyzed (Participants) | 1 | 4 | 8 | 7 | 8 | 33
  2.75 Hours Post Randomization/Treatment | 98.0 (0) | 94.5 (1.29) | 94.1 (3.64) | 94.7 (2.63) | 92.8 (4.13) | 93.5 (2.99)
  3.00 Hours Post Randomization: number analyzed (Participants) | 0 | 4 | 8 | 8 | 8 | 33
  3.00 Hours Post Randomization |  | 93.5 (5.45) | 95.0 (2.45) | 95.4 (3.46) | 94.9 (3.36) | 93.9 (2.52)

4. Primary Outcome: Serum Electrolytes
Time Frame: 24 Hours Post Randomization
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Aerosolized Lucinactant (High Dose): 75 mg TPL/kg of Lucinactant for inhalation with nCPAP
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (High Dose) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
mEq/L
  Sodium | 140 (3.7) | 137 (4.0) | 139 (4.2) | 140 (4.9) | 137 (4.3) | 139 (3.3)
  Chloride: number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 39
  Chloride | 108 (3.0) | 107 (4.2) | 107 (6.6) | 107 (6.3) | 105 (4.5) | 108 (3.5)
  Potassium | 3.86 (0.262) | 4.66 (1.235) | 3.86 (0.453) | 4.46 (1.029) | 4.09 (0.993) | 4.47 (1.082)
  Total Carbon Dioxide: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 39
  Total Carbon Dioxide | 20.8 (1.83) | 21.3 (2.12) | 22.0 (1.60) | 24.5 (7.50) | 21.9 (1.89) | 21.7 (3.12)

5. Secondary Outcome: PCO2
Description: Arterial carbon dioxide
Time Frame: Within 3 Hours of Randomization
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of arterial carbon dioxide
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (75 mg/kg) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
percentage of arterial carbon dioxide
  At Randomization: number analyzed (Participants) | 1 | 3 | 7 | 6 | 6 | 20
  At Randomization | 58.0 (0.00) | 54.3 (8.96) | 47.1 (8.32) | 49.6 (10.73) | 57.4 (10.28) | 49.2 (12.10)
  At Initiation of Treatment: number analyzed (Participants) | 3 | 6 | 6 | 7 | 8 | 0
  At Initiation of Treatment | 29.0 (1.73) | 53.0 (9.34) | 52.3 (11.34) | 46.6 (11.35) | 57.5 (6.79) |
  15 Minutes Post Randomization/Treatment: number analyzed (Participants) | 0 | 6 | 7 | 7 | 8 | 22
  15 Minutes Post Randomization/Treatment |  | 50.1 (10.42) | 53.1 (16.03) | 45.6 (9.81) | 53.0 (8.35) | 49.5 (10.82)
  30 Minutes Post Randomization/Treatment: number analyzed (Participants) | 2 | 5 | 8 | 7 | 8 | 20
  30 Minutes Post Randomization/Treatment | 38.0 (12.73) | 53.1 (8.37) | 48.4 (12.13) | 44.7 (9.62) | 55.0 (4.20) | 48.1 (9.84)
  45 Minutes Post Randomization/Treatment: number analyzed (Participants) | 1 | 6 | 7 | 7 | 8 | 23
  45 Minutes Post Randomization/Treatment | 32.0 (0.00) | 50.3 (7.94) | 46.2 (9.41) | 45.1 (10.27) | 52.6 (6.68) | 47.1 (9.67)
  60 Minutes Post Randomization/Treatment: number analyzed (Participants) | 1 | 6 | 7 | 7 | 8 | 25
  60 Minutes Post Randomization/Treatment | 39.0 (0.00) | 49.7 (9.62) | 47.3 (11.53) | 46.2 (10.02) | 51.6 (7.62) | 47.8 (7.85)
  1.25 Hours Post Randomization/Treatment: number analyzed (Participants) | 0 | 6 | 7 | 7 | 8 | 25
  1.25 Hours Post Randomization/Treatment |  | 50.5 (9.72) | 46.8 (10.55) | 44.3 (10.74) | 52.7 (8.70) | 47.5 (8.65)
  1.50 Hours Post Randomization/Treatment: number analyzed (Participants) | 0 | 6 | 6 | 7 | 7 | 24
  1.50 Hours Post Randomization/Treatment |  | 47.5 (9.62) | 46.0 (11.32) | 45.6 (10.40) | 52.3 (10.64) | 47.9 (7.12)
  1.75 Hours Post Randomization/Treatment: number analyzed (Participants) | 1 | 6 | 6 | 7 | 8 | 22
  1.75 Hours Post Randomization/Treatment | 48.0 (0.00) | 45.7 (8.44) | 44.6 (9.10) | 46.7 (8.73) | 51.8 (7.80) | 48.1 (6.46)
  2.00 Hours Post Randomization/Treatment: number analyzed (Participants) | 1 | 5 | 8 | 7 | 8 | 22
  2.00 Hours Post Randomization/Treatment | 30.0 (0.00) | 46.6 (7.72) | 45.3 (8.89) | 46.9 (9.24) | 51.0 (8.73) | 48.8 (5.90)
  2.25 Hours Post Randomization/Treatment: number analyzed (Participants) | 2 | 5 | 7 | 7 | 7 | 24
  2.25 Hours Post Randomization/Treatment | 33.5 (10.61) | 45.4 (8.49) | 47.3 (5.94) | 45.6 (8.00) | 52.9 (8.52) | 48.2 (8.56)
  2.50 Hours Post Randomization/Treatment: number analyzed (Participants) | 1 | 5 | 7 | 7 | 8 | 24
  2.50 Hours Post Randomization/Treatment | 36.0 (0.00) | 45.6 (7.20) | 42.4 (10.95) | 46.3 (10.00) | 52.0 (8.09) | 48.2 (7.64)
  2.75 Hours Post Randomization/Treatment: number analyzed (Participants) | 1 | 5 | 6 | 7 | 8 | 25
  2.75 Hours Post Randomization/Treatment | 37.0 (0.00) | 44.2 (5.02) | 46.0 (4.73) | 46.8 (8.29) | 49.9 (7.83) | 47.3 (6.94)
  3.00 Hours Post Randomization/Treatment: number analyzed (Participants) | 0 | 5 | 6 | 7 | 8 | 26
  3.00 Hours Post Randomization/Treatment |  | 45.6 (6.54) | 45.2 (5.19) | 45.9 (8.06) | 51.6 (7.09) | 46.3 (7.01)

ADVERSE EVENTS:
Time Frame: From enrollment to 36 weeks post-menstrual age (PMA). As infants are enrolled at a gestational age of 29 to 34 weeks PMA, this represents a period of 2 to 7 weeks.
Arm/Group | Aerolized Lucinactant (25 mg/kg) | Aerosolized Lucinactant (50 mg/kg) | Aerosolized Lucinactant (75 mg/kg) | Aerosolized Lucinactant (100 mg/kg) | Aerosolized Lucinactant (150 mg/kg) | nCPAP Alone
Serious Adverse Events (participants affected / at risk) | 2/8 | 3/8 | 2/8 | 3/8 | 3/8 | 7/40
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 7/8 | 8/8 | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerolized Lucinactant (25 mg/kg) (N=8) | Aerosolized Lucinactant (50 mg/kg) (N=8) | Aerosolized Lucinactant (75 mg/kg) (N=8) | Aerosolized Lucinactant (100 mg/kg) (N=8) | Aerosolized Lucinactant (150 mg/kg) (N=8) | nCPAP Alone (N=40)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 4 (5)
Necrotising Enterocolitis Neonatal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cadio-respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnoea Neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerolized Lucinactant (25 mg/kg) (N=8) | Aerosolized Lucinactant (50 mg/kg) (N=8) | Aerosolized Lucinactant (75 mg/kg) (N=8) | Aerosolized Lucinactant (100 mg/kg) (N=8) | Aerosolized Lucinactant (150 mg/kg) (N=8) | nCPAP Alone (N=40)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia Neonatal (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 15 (15)
Acrochordon (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alveolar Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apnoea Neonatal (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (4) | 2 (2) | 4 (4) | 23 (23)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Urea Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 6 (6)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary Dysplasia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive Protein Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac Murmur (Investigations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 6 (7)
Catheter Site Infection (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CNS Ventriculitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital Choroid Plexus Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital Naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 6 (6) | 2 (2) | 2 (2) | 5 (6) | 14 (15)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 16 (17)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteral Feeding Intolerance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema of Eyelid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperchloraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia Neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infantile Spasms (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Site Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intraventricular Haemorrhage Neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 8 (8) | 7 (7) | 5 (5) | 7 (8) | 30 (31)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 11 (11)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neonatal Respiratory Distress Syndrome (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Neonatal Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema Genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Pectus Excavatum (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Periorbital Oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Persistent Foetal Circulation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Poor Peripheral Circulation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Artery Stenosis Congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Interstitial Emphysema Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Pneumatocele (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal Anomaly Congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Ventricular Systolic Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis Neonatal (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient Tachypnoea of the Newborn (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (2) | 3 (3)
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days